CLINICAL TRIAL: NCT00113893
Title: A Randomized, MultiCenter, Open-Label, Modified Dose-Ascension, Parallel Study of the Safety, Tolerability, and Efficacy of Oral SCIO-469 in Patients With Myelodysplastic Syndromes
Brief Title: SCIO-469: Open-Label Study for Patients With Myelodysplastic Syndromes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005179; NCT00744432 (obsolete NCT alias)
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Bone Marrow Diseases; Myelodysplastic Syndromes; Hematologic Diseases; Bone Marrow Neoplasms
Keywords: Myelodysplastic syndromes; p38 MAP kinase; Bone marrow diseases; SCIO-469
MeSH Terms: conditions — Bone Marrow Diseases; Myelodysplastic Syndromes; Hematologic Diseases; Bone Marrow Neoplasms | interventions — SCIO-469

ARMS (4):
- Scio-469 30 Milligram (mg) (Experimental): SCIO-469 tablet will be administered orally at a dose of 30 mg thrice daily (90 mg per day) for 16 weeks. Participants with hematologic improvement at Week 16 and as per Investigator's discretion on clinical benefit from treatment will continue the treatment for additional 36 weeks.
  Interventions: Drug: SCIO-469
- Scio-469 60 mg (Experimental): SCIO-469 tablet will be administered orally at a dose of 60 mg thrice daily (180 mg per day) for 16 weeks. Participants with hematologic improvement at Week 16 and as per Investigator's discretion on clinical benefit from treatment will continue the treatment for additional 36 weeks.
  Interventions: Drug: SCIO-469
- Scio-469 90 mg (Experimental): SCIO-469 tablet will be administered orally at a dose of 90 mg thrice daily (270 mg per day) for 16 weeks. Participants with hematologic improvement at Week 16 and as per Investigator's discretion on clinical benefit from treatment will continue the treatment for additional 36 weeks.
  Interventions: Drug: SCIO-469
- Scio-469 120 mg (Experimental): SCIO-469 tablet will be administered orally at a dose of 120 mg thrice daily (360 mg per day) for 16 weeks. Participants with hematologic improvement at Week 16 and as per Investigator's discretion on clinical benefit from treatment will continue the treatment for additional 36 weeks.
  Interventions: Drug: SCIO-469

INTERVENTIONS:
Drug: SCIO-469 — SCIO-469 tablet will be administered orally at a dose of 30 mg thrice daily (90 mg per day) for 16 weeks. Participants with hematologic improvement at Week 16 and as per Investigator's discretion on clinical benefit from treatment will continue the treatment for additional 36 weeks.
  Arms: Scio-469 30 Milligram (mg)
Drug: SCIO-469 — SCIO-469 tablet will be administered orally at a dose of 60 mg thrice daily (180 mg per day) for 16 weeks. Participants with hematologic improvement at Week 16 and as per Investigator's discretion on clinical benefit from treatment will continue the treatment for additional 36 weeks.
  Arms: Scio-469 60 mg
Drug: SCIO-469 — SCIO-469 tablet will be administered orally at a dose of 90 mg thrice daily (270 mg per day) for 16 weeks. Participants with hematologic improvement at Week 16 and as per Investigator's discretion on clinical benefit from treatment will continue the treatment for additional 36 weeks.
  Arms: Scio-469 90 mg
Drug: SCIO-469 — SCIO-469 tablet will be administered orally at a dose of 120 mg thrice daily (360 mg per day) for 16 weeks. Participants with hematologic improvement at Week 16 and as per Investigator's discretion on clinical benefit from treatment will continue the treatment for additional 36 weeks.
  Arms: Scio-469 120 mg

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of oral SCIO-469 in patients with myelodysplastic syndromes. SCIO-469 belongs to a new class of treatments that inhibit expression and activity of cytokines that play a role in the progression of MDS.

DETAILED DESCRIPTION:
SCIO-469 belongs to a new class of treatment that inhibits p38 MAP kinase. p38 MAPK activation controls the production of TNF-a, VEGF, and IL-1b. As an inhibitor of p38 MAPK, SCIO-469 blocks the synthesis of these molecules, as well as TNF-a activity. This randomized, open-label, modified dose-ascension study is designed to assess the safety, tolerability, and efficacy of oral SCIO-469 in the treatment of patients with MDS. This patient group was selected because of the inhibitory effect of SCIO-469 on the expression and activity of cytokines that play a role in the progression of MDS. The treatment arms will be 30, 60 , 90, or 120 mg tid with 15 subjects per arm (total of 60 subjects) and each arm may expand to 25 subjects per arm (maximum total of 100 subjects). Initially, subjects will be randomly assigned to one of the lowest two treatment arms (30 mg tid or 60 mg tid). When 6 subjects per arm (at least 12 subjects total) have received study drug for at least 4 weeks, predefined criteria will be used to determine whether to open randomization into the third arm (i.e., 90 mg tid). The criteria will be based on the number of subjects who have had to suspend study drug due to drug-related toxicity. The 120-mg tid arm will be open for enrollment after 15 subjects have been enrolled into each of the first three treatment arms; the decision to open enrollment will be similar to the criteria used to open the third arm. Subjects will be evaluated at least monthly for safety and some efficacy measurements (AE reporting, safety labs and vitals). Subjects will receive study drug for 16 weeks. Subjects who demonstrate hematologic improvement (erythroid, platelet, or neutrophil response by IWG criteria) at week 16 will be eligible to continue treatment at the same dose of study drug for up to 36 additional weeks (52 weeks of total drug exposure). Subjects who do not meet the IWG criteria for hematologic improvement at week 16 but who, in the judgment of the investigator, experience clinical benefit may also receive up to 36 additional weeks of treatment. The same judgments for treatment extensions of additional 26 weeks in responding subjects will be made at 52 weeks and 78 weeks; maximum total drug exposure will be 104 weeks. All subjects will be followed for 4 weeks after the last study drug treatment for safety assessments or until resolution of Grade 3 or greater treatment-related toxicity as defined by NCI CTCAE (v. 3.0).

Oral SCIO-469 given for 16 weeks to patients with MDS. Subjects will receive a total daily dose of SCIO-469 of 90 mg, 180 mg, 270 mg, or 360 mg. The treatment arms will be 30-mg tablet tid, 60-mg tablet tid, 90-mg tablet tid, or 120 mg (i.e., two 60-mg tablets) tid with 15 subjects per arm (total of 60 subjects). Responding subjects may dose for up to 104 weeks total drug exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of low/intermediate-1 MDS (for at least 12 weeks)
* Patients with anemia (average Hemoglobin < 10 g/dL or > or = to 4 units of Red Blood Cell counts in the last 8 weeks)
* Patients who have failed prior erythropoietin treatment
* Patients with an ECOG (Eastern Collaborative Oncology Group) score of 0, 1 or 2

Exclusion Criteria:

* Patients with a International Prognostic Scoring System risk category high/intermediate-2
* Patients with treatment-related MDS associated with radiation, chemotherapy, and/or autologous transplant
* Patients with myelosclerosis (or myelofibrosis) occupying > 30 % marrow space
* Patients who have received decitabine (DacogenTM) for MDS
* Patients who have received lenalidomide (RevlimidTM), steroids, erythropoietin, hydroxyurea, or growth factors within 4 weeks before study drug administration
* Patients who have received thalidomide within 8 weeks before study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Major or Minor Erythroid Response (Hematological Improvement - Erythroid [HI-E]) | Week 16
  Improvement in Erythroid (HI-E) lineage will be assessed as per International Working Group (IWG) criteria. HI-E major response is defined as greater than 2.0 gram per deciliter g/dL increase in hemoglobin for red blood cell (RBC) transfusion-dependent participants, transfusion independence. HI-E minor response is defined as 1.0 to 2.0 g/dL increase in hemoglobin for RBC transfusion-dependent participants and 50 percent decrease in transfusion requirements.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Major or Minor Neutrophil Response (HI-N) | Week 16
  Major or minor neutrophils response is Hematologic Improvement in Neutrophil (HI-N) lineage. It will be assessed as per International Working Group (IWG) criteria. HI-N major response is defined as for participants with pre-treatment Absolute Neutrophil Count (ANC) less than 1500 per micro (l), at least 100 percent increase or an absolute increase more than 500 per micro l, whichever is greater. HI-N minor response defined as for participants with pre-treatment ANC less than 1500 per micro l, ANC increase of at least 100 percent, but with absolute increase less than 500 per micro l.
Percentage of Participants Achieving Major or Minor Platelet Response (HI-P) | Week 16
  Major or minor neutrophils response is Hematologic Improvement in Platelets (HI-P) lineage. It will be assessed as per International Working Group (IWG) criteria. HI-P major response is defined as for participants with pre-treatment platelet count less than 100,000 per micro liter (l ), an absolute increase of 30,000 micro l or more. HI-P minor response defined as for participants with pre-treatment platelet count less than 100,000 per micro l, a 50 percent or more increase in platelet count with net increase greater than 10,000 per micro l but less than 30,000 per micro l.
Percentage of Participants Achieving Complete or Partial Bone Marrow (BM) Response | Week 16
  Bone marrow response will be assessed as per the IWG criteria. Bone marrow response categories are: complete remission and partial remission. Complete remission is defined as normal bone marrow morphology (less than 5 percent myeloblasts with no cytologic dysplasia). Partial remission is defined as (must last at least 8 weeks) blasts decreased by 50 percent or more over pre-treatment, or a less advanced Myelodysplastic syndrome (MDS) French-American and British (FAB) classification than pre-treatment
Percentage of Participants Achieving Major or Minor Cytogenetic Response | Week 16
  Cytogenetic response will be assessed as per IWG criteria. Major response is defined as no detectable cytogenetic abnormality, if pre-existing abnormality was present. Minor response is defined as greater than percent 50 reductions in abnormal metaphases.

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.